CLINICAL TRIAL: NCT01418534
Title: An Open Label, Randomized, Two Treatment, Two Sequence, Two Period, Cross-over, Single-dose Comparative Oral Bioavailability Study of Isosorbide Mononitrate 120 mg ER Tablets (Test) of Torrent Pharmaceuticals Ltd., India and Isosorbide Mononitrate 120 mg ER Tablets (Reference) of Kremers Urban, USA in Healthy, Adult, Male, Human Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Torrent Pharmaceutical Limited's ISMN 120 mg ER Tablets Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Chief Investigator, Torrent Pharmaceuticals Limited
Other Study IDs: 179/09
Record Dates: First submitted 2011-08-11; First posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-08

CONDITIONS: Healthy

INTERVENTIONS:
Drug: Torrent's Isosorbide Mononitrate 120 mg ER Tablets

SUMMARY:
Objective:

to compare the single dose bioavailability of Torrent's Isosorbide Mononitrate 120 mg ER Tablets (Test) and Isosorbide Mononitrate 120 mg ER Tablets (Reference) of Kremers Urban, USA. Dosing periods were separated by a washout period of 8 days.

Study Design:

randomized, two-way crossover, single-dose, open-label study in healthy human adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy males within the age range of 18 to 55 years.
* A body mass index within 18-25 Kg/m2.
* Given written informed consent to participate in the study.
* Absence of diseases markers of HIV 1 & 2, Hepatitis B & C virus and RPR.
* Absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history and physical examination during the screening.
* A normal 12-lead ECG.
* A normal chest X-Ray.
* Comprehension of the nature and purpose of the study and compliance with the requirements of the entire protocol.
* No history or no evidence of hypersensitivity or idiosyncratic reactions to other nitrates or nitrites.
* No history of allergic rash.
* No history of significant systemic diseases.
* No history of psychiatric disorders or addiction to any recreational drug or drug dependence.
* No donation of blood within 56 days prior to study check-in.
* No participation in any clinical study within the past 56 days.
* No receipt of any prescription drugs or OTC products, with in two weeks prior to study check-in.
* No history of dehydration from diarrhea, vomiting or any other reason within a period of 24 hours prior to study check-in.
* No family history of neurological disorders.
* Not consumed alcohol and xanthine containing food and beverages, cigarettes and tobacco products, for at-list 48 hours, prior to study check-in.
* Negative results for drugs of abuse in urine and alcohol breath analysis during check-in of each period.
* Not consumed grape fruit juice within the 48 hours prior to study check-in.

Exclusion Criteria:

* Blood pressure Systolic> 140 mm Hg and < 110 mm Hg Diastolic< 70 mm Hg > 90 mm Hg
* History of seizures
* History of alcohol consumption for more than 2 units/day.
* High caffeine or tobacco consumption
* History of difficulty with donating blood or difficulty in accessibility of veins.
* Any unusual or abnormal diet, for whatever reason e.g. fasting due to religious reasons.
* Used any pharmacological agents known to significantly induce or inhibit drug metabolizing enzymes within 14 days of the start of the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult

PRIMARY OUTCOMES:
bioequivalence based on Composite of Pharmacokinetics
  bioequivalence; 90% geometric confidence interval of the ratio of least-squares means of the test to reference product should be within 80.00% - 125.00% for AUC-unf, AUCo-t and Cmax.

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Trident Life sciences Limited, Hyderabad, Andhra Pradesh
  - Trident Life Sciences Limited, Hydrabad, Andhra Pradesh